CLINICAL TRIAL: NCT06265246
Title: The Effects of Milk and Yogurt Supplementation on Bone Health, Body Composition, and Gut Microbiota in Canadian Young Adults: A Randomized Controlled Trial
Brief Title: Impact of Milk and Yogurt Supplementation on Bone Health, Body Composition, and Gut Microbiota in Canadian Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Dairy Farmers of Canada (Other); Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Hassanali Vatanparast, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104993
Record Dates: First submitted 2024-02-01; First posted 2024-02-20 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Osteoporosis; Obesity
Keywords: probiotics; cultured milk products; milk; osteoporosis; obesity; gastrointestinal microbiome; body composition; yogurt
MeSH Terms: conditions — Osteoporosis; Obesity | interventions — Milk; Yogurt

STUDY DESIGN:
Intervention Model Description: In this 24-month randomized controlled trial, the investigators will follow the Consolidated Standards of Reporting Trials (CONSORT) guidelines. Ninety-nine free-living adults aged 19-30 years with low dietary calcium intake will be randomly assigned to one of the following three intervention arms.
  1. Habitual diet (control) (n=33)
  2. Habitual diet + 1.5 servings of milk providing approx. 500 mg Ca/day (either 1% fat milk, or 2% fat milk) (n=33)
  3. Habitual diet + 2 servings of yogurt providing approx. 500 mg Ca/day (either 1% fat plain yogurt, 2% fat plain yogurt, 1% fat flavoured yogurt, 2% fat flavoured yogurt) (n=33)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Habitual Diet (Control) (No Intervention): 33 participants in this arm will continue to take their usual diet without any intervention.
- Habitual Diet + 1.5 Servings of Milk (Experimental)
  Interventions: Other: Habitual Diet + Milk
- Habitual Diet + 2 Servings of Yogurt (Experimental)
  Interventions: Other: Habitual Diet + Yogurt

INTERVENTIONS:
Other: Habitual Diet + Milk — 1.5 servings of milk [providing approx. 500 mg Ca/day] per day (either 1% fat milk, or 2% fat milk)
  Arms: Habitual Diet + 1.5 Servings of Milk
Other: Habitual Diet + Yogurt — 2 servings of yogurt [providing approx. 500 mg Ca/day] per day (either 1% fat plain yogurt, 2% fat plain yogurt, 1% fat flavoured yogurt, 2% fat flavoured yogurt)
  Arms: Habitual Diet + 2 Servings of Yogurt

SUMMARY:
Milk and dairy products contain significant amounts of nutrients that contribute to optimal health - nutrients like calcium, vitamin D, and high-quality protein. Fermented milk products or fermented dairy products are dairy foods that have been fermented with certain bacteria. Yogurt is a fermented dairy product containing millions of beneficial bacteria. In this study, the invesgitagtors will look at the effect of milk (a non-fermented dairy product) and yogurt (a fermented dairy product) supplementation on bone health and the amount of fat and muscle mass in Canadian young adults over a 24-month period. While dairy products contain significant amounts of nutrients, the scientific community does not know the impact of long-term supplementation of fermented (i.e., yogurt) or non-fermented (i.e., milk) dairy food on bone health and the amount of fat and muscle mass in young adults. To fill this knowledge gap, the investigators will recruit participants with low calcium intake and assign them to three different groups: 1) milk (intervention) group; 2) yogurt (intervention) group; and 3) control group. The investigators will ask the participants in the milk group to drink 1.5 servings (375 mL) of milk per day for 24 months. Participants in the yogurt group will consume 2 servings (350 g) of yogurt per day for 24 months. Those in the control group will continue their usual diets. Using a randomized controlled trial design, the investigators will measure bone health parameters, hormonal indices related to bone metabolism, body composition (e.g., muscle mass, fat mass), and the number and composition of bacteria living in the gastrointestinal (GI) tract. The hypothesis is that supplementation with yogurt will have more positive effects on bone health indices, particularly femoral neck BMD as the primary outcome, than milk in Canadian adults aged 19-30 years. The secondary hypothesis is that supplementation with yogurt, as a fermented milk product, will have a more beneficial effect than milk on body composition measures. The data will provide valuable information for developing targeted health initiatives and marketing strategies regarding the benefits of fermented and non-fermented dairy product consumption.

DETAILED DESCRIPTION:
The overarching goal of this project is to determine the role of milk and yogurt supplementation on bone health and body composition in Canadian adults aged 19 to 30 years. Both the prevalence of obesity and osteoporosis among Canadians reflect a public health concern. According to data from 2018, 27% of Canadians aged 18 and older were classified as obese, and 36% were classified as overweight. Data from 2016 revealed a diagnosis of osteoporosis for 12% of Canadians. Consumption of milk and milk products play a role in bone homeostasis over the life course but most of the research has focused on children or older adults. Dairy product intake is associated with lower body weight or body fat. However, Canadian cross-sectional data shows a decline in the consumption of dairy products among all ages from 2004 to 2015. The overall impact of dairy consumption trends is reflected in the prevalence of calcium inadequacy among Canadians. Previous studies suggest that dairy products may positively influence bone homeostasis and body composition through various mechanisms involving key nutrients and the contribution of probiotics. Young adults are in a transitional period and thus at a critical point for developing healthy lifestyle habits that support optimal body composition and maintenance of peak bone mineral density. Further, as fermented milk products contain many beneficial nutrients, determining the specific role probiotics play is difficult to define. The research will build on previous studies with a specific focus on addressing current knowledge gaps on the health impacts of young adults and the comparison between milk and yogurt.

The specific objectives of the research are:

1. To examine the effects of milk and yogurt supplementation on bone mineral density (BMD), bone mineral content (BMC), bone structure, and bone geometry of Canadian adults aged 19-30 years.
2. To examine the effects of milk and yogurt supplementation on hormonal indices (parathyroid hormone, Insulin-like growth factor 1, 25-hydroxyvitamin D) related to bone metabolism in Canadian adults aged 19 to 30.
3. To examine the effects of milk and yogurt supplementation on biochemical indices of bone turnover (Procollagen type 1 N-propeptide, Osteocalcin, Bone alkaline phosphatase, N-terminal telopeptide of type I collagen, C-terminal telopeptide of type 1 collagen) in Canadian adults aged 19-30.
4. To examine the effects of milk and fermented milk product supplementation on body composition (bone-free lean tissue mass, total body fat mass, abdominal fat mass, percent total body fat) of Canadian adults aged 19 to 30.
5. To examine the effects of milk and fermented milk product supplementation on gut microbiota of Canadian adults aged 19 to 30

ELIGIBILITY:
Inclusion Criteria:

* 19-30 years old
* Dietary calcium intake below 1000mg/ day
* living in the Saskatoon area (Saskatchewan, Canada)

Exclusion Criteria:

* Calcium intake from both food and supplement above the estimated average requirement (EAR) for adults aged 19-30 years (>800 mg/day)
* Total dairy intake of more than 1 serving per day
* Body mass index greater than to 30 kg/m2
* Medical history of metabolic bone, liver, endocrine, connective tissue, and respiratory diseases, thyroid disorders, or cancer
* Diagnosed cases with secondary osteoporosis due to hypoparathyroidism
* Hormonal disorders or disturbances
* Taking medications known to influence bone mass and density (e.g., steroids, diuretics, heparin, and cancer drugs)
* Cow's milk allergy
* Pregnant or lactating women, or those planning to conceive during the duration of the trial

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Femoral neck bone mineral density | Baseline, month 12, month 24
  Measurement will be done via Dual Energy X-ray Absorptiometry.

SECONDARY OUTCOMES:
Bone mineral density (total hip, lumbar spine, whole body) | Baseline, month 12, month 24
  Measurement will be done via Dual Energy X-ray Absorptiometry.
Bone mineral content (total hip, femoral neck, lumbar spine, whole body) | Baseline, month 12, month 24
  Measurement will be done via Dual Energy X-ray Absorptiometry.

OTHER OUTCOMES:
Bone structure | Baseline, month 12, month 24
  Measurement via HR-pQCT scan at distal radius and tibia
Bone geometry | Baseline, month 12, month 24
  Measurement via HR-pQCT scan at distal radius and tibia
Serum bone alkaline phosphatase (biochemical indices of bone turnover) | Baseline, month 12, month 24
  Fasting blood sample will be collected from each participant between 8 a.m. and 10 a.m. after an overnight fast of 12 hours with no heavy exercise/workouts 48 hours prior to blood collection into 2 x 4ml serum separating tubes (SST) for the analysis of all serum measures.
Serum osteocalcin (biochemical indices of bone turnover) | Baseline, month 12, month 24
  Fasting blood sample will be collected from each participant between 8 a.m. and 10 a.m. after an overnight fast of 12 hours with no heavy exercise/workouts 48 hours prior to blood collection into 2 x 4ml serum separating tubes (SST) for the analysis of all serum measures.
Serum procollagen type 1 N-propeptide (biochemical indices of bone turnover) | Baseline, month 12, month 24
  Fasting blood sample will be collected from each participant between 8 a.m. and 10 a.m. after an overnight fast of 12 hours with no heavy exercise/workouts 48 hours prior to blood collection into 2 x 4ml serum separating tubes (SST) for the ananalysis of all serum measures.
Serum N-terminal telopeptide of type 1 collagen (biochemical indices of bone turnover) | Baseline, month 12, month 24
  Fasting blood sample will be collected from each participant between 8 a.m. and 10 a.m. after an overnight fast of 12 hours with no heavy exercise/workouts 48 hours prior to blood collection into 2 x 4ml serum separating tubes (SST) for the analysis of all serum measures.
Serum C-terminal telopeptide of type 1 collagen (biochemical indices of bone turnover) | Baseline, month 12, month 24
  Fasting blood sample will be collected from each participant between 8 a.m. and 10 a.m. after an overnight fast of 12 hours with no heavy exercise/workouts 48 hours prior to blood collection into 2 x 4ml serum separating tubes (SST) for the aanalysis of all serum measures.
Serum PTH (hormonal indices related to bone metabolism) | Baseline, month 12, month 24
  Fasting blood samples will be collected from each participant between 8 a.m. and 10 a.m. after an overnight fast of 12 hours with no heavy exercise/workouts 48 hours prior to blood collection for the analysis of all serum measures.
Serum 25(OH)D (hormonal indices related to bone metabolism) | Baseline, month 12, month 24
  Fasting blood samples will be collected from each participant between 8 a.m. and 10 a.m. after an overnight fast of 12 hours with no heavy exercise/workouts 48 hours prior to blood collection for the analysis of all serum measures.
Serum IGF-1 (hormonal indices related to bone metabolism) | Baseline, month 12, month 24
  Fasting blood samples will be collected from each participant between 8 a.m. and 10 a.m. after an overnight fast of 12 hours with no heavy exercise/workouts 48 hours prior to blood collection for the analysis of all serum measures.
Saliva IGF-1 (hormonal indices related to bone metabolism) | Baseline, month 12, month 24
  Saliva samples will be collected from each participant for analysis of salivary IGF-1 and comparison to serum IGF-1.
Fat mass and lean mass | Baseline, month 12, month 24
  Measurement via Dual Energy X-ray Absorptiometry.
Height | Baseline, month 12, month 24
  Height (cm) in standing position will be measured to the nearest 0.1 cm by a wall-mounted stadiometer.
Weight | Baseline, month 12, month 24
  For weight measurements, participants will be asked to wear light clothes and remove their shoes and jewelry and then stand on the SECA electronic scale to measure the weight to the nearest 0.01 kg.
Gut microbiota via general lactobacillus and bifdobacterium | Baseline, month 12, month 24
  Stool samples will be collected using DNAgenotek Omnigene sample collection kits and the total DNA of gut microbiomes from fecal material will be extracted using QIAamp PowerFecal Pro DNA Kit (Cat No. 51804), following manufacturer's instructions
Dietary assessment | Baseline, month 6, month 12, month 18, month 24
  Dietary intake will be assessed using serial 24-hour dietary recalls. Dietary data will be collected in person at baseline, 12 months, and 24 months and via telephone at 6 months and 18 months. The mean of three 24-h recalls at each time point will provide an estimation of the usual intake.
Physical activity | Baseline, month 6, month 12, month 18, month 24
  Physical activity will be captured using the Physical Activity Adult Questionnaire (PAAQ) to include transportation, recreational, and occupational or household physical activity in the last 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Vatanparast, MD, PhD, Principal Investigator — University of Saskatchewan; Phil Chilibeck, PhD, Principal Investigator — University of Saskatchewan; Sandra Clarke, Principal Investigator — Agriculture and Agri-Food Canada
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No